CLINICAL TRIAL: NCT06924359
Title: Multimodal Ophthalmic Imaging and Plasma Biomarkers for the Early Detection of Alzheimer's Disease
Acronym: MOIPAD
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AD-BIOPR-001
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease (AD)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Different stages of Alzheimer's disease
  Interventions: Diagnostic Test: Multimodal Ophthalmic Imaging and plasma biomarker

INTERVENTIONS:
Diagnostic Test: Multimodal Ophthalmic Imaging and plasma biomarker — Multimodal Ophthalmic Imaging and plasma biomarkers (Aβ42/40, p-tau181, p-tau217, NfL and GFAP）.

SUMMARY:
With the accelerating global aging population, dementia has become a pressing worldwide issue. This project aims to identify specific plasma biomarkers and ocular indicators for the early detection of Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥ 50 years;
* Participants diagnosed with Alzheimer's Disease (AD), mild cognitive decline (MCI), subjective cognitive decline (SCD), or cognitively normal (CN);
* Signed informed consent form

Exclusion Criteria:

* Presence of other neurological disorders and systemic diseases that may cause cognitive impairment;
* Inability to cooperate with cognitive assessments;
* Refusal to undergo blood sampling.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: AD, MCI, SCD and CN
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Differences in Multimodal Ophthalmic Imaging parameter values among groups | Baseline

SECONDARY OUTCOMES:
Concentration difference of plasma biomarkers (Aβ42/40, p - tau181, p - tau217, NfL and GFAP） among groups | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No